CLINICAL TRIAL: NCT06818760
Title: Single Center Pilot Study of Remote Monitoring in Pregnant Women With Congenital Heart Disease Using Wrist Wearables
Brief Title: Remote Monitoring in Pregnant Women With Congenital Heart Disease Using Wrist Wearables
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-1183
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease; Congenital Vascular Disorder; Congenital Cardiomyopathy; Pregnancy Related
MeSH Terms: conditions — Heart Defects, Congenital; Cardiomyopathy, infantile histiocytoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Masimo Smart Wristband: Masimo Smart Wristband continuous ambulatory monitoring
  Interventions: Diagnostic Test: Masimo Smart Wristband

INTERVENTIONS:
Diagnostic Test: Masimo Smart Wristband — Continuous wear of Masimo Smart Wristband

SUMMARY:
Congenital heart disease (CHD) includes a wide variety of types of disease, including congenital abnormalities of the heart valves. This can range from bicuspid aortic valve and other aortic valve deformities to more complex disease such as tetralogy of Fallot.

For many kinds of CHD, the optimal timing of interventions remains unclear. For instance, in tetralogy of Fallot, there is still equipoise about when to offer pulmonary valve replacement (PVR), while in aortic regurgitation, some patients can remain stable for many years.

The primary focus of this study is to use continuous physiologic data (CPD), obtained using wearable biosensors (a type of biometric monitoring technology), to develop improved biomarkers of disease progression and prognosis from patients with congenital heart disease (CHD) who are pregnant while they are at home as well as looking at patients' experience and interaction with wearable biosensor technology at home.

DETAILED DESCRIPTION:
Maternal cardiovascular disease (MCD) remains the leading cause of death in pregnant women, especially in the United States, where heart disease is on the rise. The worse outcomes disproportionately affect disadvantaged populations, including those with poor access to healthcare, and ethnic minorities. Reducing maternal mortality is a World Health Organization global health goal, and multiple efforts have been initiated to both study maternal cardiac disease as well as reduce morbidity and mortality. At least half of serious cardiac complications can be prevented with closer monitoring and adequate care. A multidisciplinary approach using the Cardio-obstetrics clinic model has been shown to improve outcomes in women with cardiovascular disease, but successful efforts have been limited to comprehensive care centers in larger cities. Over the past decades, there have also been advances in the risk assessment for pregnant women with cardiac disease, but all risk models have not been as accurate in validation models and further research is warranted.

Hemodynamic changes of pregnancy, during labor, and in the early postpartum period include a decrease in systemic vascular resistance (SVR) and increases in blood volume and heart rate, all resulting in increased cardiac output (CO). There is also an associated increase in ventricular muscle mass and end diastolic volumes with improved systolic function, but without a pathologic increase in end-diastolic pressures. Such hemodynamic and anatomic alterations can exacerbate underlying cardiac disease, as well as uncover previously unrecognized cardiovascular pathology, thereby increasing the risk of cardiac complications.12 Several cardiac complications during pregnancy and in the postpartum period are due to the inapt response to pregnancy with either an inability to augment CO or inability to tolerate the increased CO. Addressing maternal cardiac complications would require earlier detection and identification of those at risk.

Wearable derived biomarkers: Physiological health parameters derived from either non-invasive monitors or wearables allow continuous tracking of such parameters in an ambulatory state:

* Pulse Oximetry (SpO2) is used to detect peripheral cyanosis, normal being >95%, and has been used to detect newborn cyanosis in children with congenital heart disease, albeit with reduced accuracy at saturations <60%.
* Respiratory rate in breaths per minute (RRp) can increase in pregnancy from 8-12 breaths per minute to 15-17 breaths per minute, but it increases to a larger extent in states of distress, infection, and cardiovascular decompensation. In one study, increased RRp, and heart rate (HR) were detected early in women that were found to have an intraamniotic infection, demonstrating the benefit of such monitors in early detection of pathology.
* Heart rate variability (HRV) measures changes in the time intervals between consecutive heartbeats and is a surrogate for neural cardiac control and the balance between the sympathetic and parasympathetic drive. Higher variability (50-100 ms) is normal with an overall decline with age. Low HRV has been shown to be a predictor of poor outcomes in patients with cardiac disease in small studies, a wearable device was used to evaluate HRV during normal pregnancy, and it was found to be overall decreased (50-70 ms), but with a dynamic burst in autonomic activity in the transition from second to third trimester
* In addition, these monitors can provide dynamic indices that include the perfusion index (Pi), which depends on the blood flow in the peripheral circulation, the cardiac output, and the vascular tone, which is calculated from the amount of light constantly absorbed by skin from non-pulsatile blood, and the variable amount of light absorbed by pulsating arterial inflow, with values ranging from 0.2%-20%, with lower percentages indicating lower perfusion state. There have been unvalidated suggestions that Pi can be used as a surrogate for CO.
* The pleth variability index (PVi), is the maximal and minimal Pi over a respiratory cycle and is also expressed in %, with a range of 9-13%. In a randomized controlled trial of intraoperative and postoperative patients, elevated PVi was used to direct fluid management by administering crystalloid infusions in PVi >13%, with appropriate fluid responsiveness. Such intervention reduced the overall fluid infused to patients, and reduced lactate levels. Elevated PVi has also been used to predict hypotension in pregnant women undergoing c-section.

Masimo® noninvasive monitors (Masimo Corp, Irvine, CA) are FDA approved for use in adults and newborns to provide real time pulse oximetry (SpO2) and heart rate. Masimo has CE mark for additional parameters which include PVR, atrial fibrillation respiratory rate per minute (RRp), heart rate variability (HRV), and PVi. Clinical studies demonstrated they are motion-tolerant, report functional oxygen saturation, and validation in low perfusion conditions. Smart wristbands are an unobtrusive, and promising novel method to monitor ambulatory health parameters throughout pregnancy. The Masimo W1® wristband is FDA approved and uses clinically tested technology in a wearable patient-friendly format. Compliance with wearable devices has been demonstrated in a small study of 20 pregnant women where it was worn approximately 6 out of 7 months, with a slight drop in adherence postpartum.

ELIGIBILITY:
Inclusion Criteria:

Women evaluated in the cardio-obstetrics clinic either prepartum, intrapartum, or postpartum with congenital heart disease.

* Congenital heart disease: Based on modified World Health Organization (mWHO) classification of maternal cardiovascular disease group ≥ II.

  * mWHO Class I include mild pulmonary stenosis, uncomplicated patent ductus arteriosus, and repaired shunts, to be excluded.
  * mWHO Class II includes unoperated atrial septal defect or ventricular septal defect and repaired tetralogy of Fallot.
  * mWHO Class II-III includes mild left ventricular impairment, valvular heart disease not in class I, repaired aortic coarctation, Marfan without aortic dilation, bicuspid aortic valve with <45 mm root, hypertrophic cardiomyopathy.
  * mWHO Class III includes systemic right ventricle, Fontan circulation, unrepaired cyanotic heart disease, Marfan with aorta 40-45 mm, bicuspid aortic valve with root 45-50 mm, other complex congenital heart disease (such as Shone complex).
  * mWHO Class IV includes Marfan with >45 mm aorta, bicuspid aortic valve with > 50 mm aorta, severe systemic ventricular dysfunction (EF<30%), severe symptomatic AS or MS, native severe coarctation, all severe pulmonary hypertension patients from any cause.
* Congenital valvular heart disease:

  * Native valvular heart disease: tricuspid, pulmonary, mitral and aortic with ≥ moderate regurgitation or stenosis by echocardiography.
  * Bioprosthetic valvular heart disease with ≥ moderate regurgitation or stenosis by echocardiography.
  * Any mechanical valve prosthesis
* Congenital Cardiomyopathy

  * Cardiomyopathy with EF < 30%
  * Cardiomyopathy with EF 30-50%
* Provide Informed consent
* Age > 18 years of age

Exclusion Criteria:

* Patients on hemodialysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women greater or equal to 18 years of age who have a congenital heart disease (congenital valvular heart disease, Native valvular heart disease, bioprosthetic valvular heart disease, any mechanical valve prosthesis and congenital cardiomyopathy with EF less then 50%) who are pregnant.
Study Population: Women greater or equal to 18 years of age who have a congenital heart disease (congenital valvular heart disease, Native valvular heart disease, bioprosthetic valvular heart disease, any mechanical valve prosthesis and congenital cardiomyopathy with EF less then 50%) who are pregnant from high risk obstetric clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
New onset atrial or ventricular arrhythmias | Up to 12 month post-partum
  New onset of atrial tachycardia, flutter or fibrillation, non-sustained VT (3 or more PVC, lasting <30 seconds), PVC burden >10% within 24 hours detected on ECG or event monitors on clinic visits or prompted by subjective palpitations, ECG or event monitor obtained routinely due to clinical suspicion of arrhythmia.

SECONDARY OUTCOMES:
Increased NT-proBNP | During the first (up to 12 weeks of gestation) and third trimester (28-40 weeks of gestation)
  Change in value of >200 pg/mL in the first and second trimester, and >150 pg/mL in the third trimester
New or worsening of biventricular dysfunction or valvular dysfunction on echocardiography | Up to 12 months post-partum
  a reduction in EF by >5%. New or worsening valvular dysfunction is defined as an increase in valve dysfunction by 1 grade of severity (mild, moderate, severe) on echocardiography.
Cardiac-related hospital or intensive care unit (ICU) admission | Up to 12 months post-partum
  Number of occurrence of cardiac-related hospital or ICU admission
Inotropic or mechanical circulatory support | Up to 12 months post-partum
  Number of occurrence of inotropic or mechanical circulatory support
Cardiac death | Up to 12 months post-partum
  Occurrence of death from cardiac-cause

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ghobrial, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States